CLINICAL TRIAL: NCT05025462
Title: Supplementation with Salmon Peptide Fraction in Overweight-Obese Men and Women: Safety, Cardiometabolic Health Effects and Mechanisms of Action
Brief Title: Salmon Peptide Fraction: Safety and Cardiometabolic Health
Acronym: SPF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, André Marette, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SPF1 2021-157
Record Dates: First submitted 2021-08-24; First posted 2021-08-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPF (Experimental): Salmon peptide fraction supplement: powder mixed in water
  Interventions: Dietary Supplement: Supplement dose 15g/d; Dietary Supplement: Supplement dose 7.5g/d
- Comparator (Active Comparator): Casein peptide fraction supplement: powder mixed in water
  Interventions: Dietary Supplement: Supplement dose 15g/d; Dietary Supplement: Supplement dose 7.5g/d

INTERVENTIONS:
Dietary Supplement: Supplement dose 15g/d — Supplementation with 15g/day of SPF or Comparator
Dietary Supplement: Supplement dose 7.5g/d — Supplementation with 7.5g/d of SPF ou comparator

SUMMARY:
The overall goal of this study is to verify the safety of 15g of salmon peptide fraction (SPF), and to test the effects on metabolic syndrome risk factors of two doses of SPF (7.5g and 15g) in overweight-obese men and women. Transcriptomic, metabolomic and metagenomic approaches will be used to study the physiological effects of SPF and to discover the potential mechanism underlying these effects.

DETAILED DESCRIPTION:
Increased fish consumption has been suggested to improve the metabolic syndrome (MetS) and to reduce the incidence of type 2 diabetes (T2D) and cardiovascular disease (CVD) in obese subjects. While it is well documented that marine long chain polyunsaturated fatty acids (n-3 PUFA) decrease CVD risk by improving the plasma lipid profile and reducing inflammation, the beneficial effects of n-3 PUFA on glucose homeostasis and insulin sensitivity in humans remains highly controversial. Animal and human studies carried out by the group of investigators over the past 20 years have shown that fish proteins can improve the plasma lipid profile, enhance insulin sensitivity and reduce obesity-linked inflammation. The investigators also reported that a salmon protein hydrolysate reduces body fat and increases insulin sensitivity via its calcitonin content and they observed that protein hydrolysates from salmon and other fish sources reduced inflammation in visceral adipose tissue in rodents. The investigators therefore decided a few years ago to focus on the identification of bioactive peptides from fish proteins to explore the potential of increasing the efficacy of fish muscle protein hydrolysates to prevent/treat the MetS. The investigators hypothesized that it was the peptides produced from gastrointestinal digestion that were responsible for the remarkable bioactive effects of fish proteins on the MetS. The investigators have also confirmed that a small peptides fraction (SPF) from salmon protein markedly reduces the development of T2D and inflammation in a high-fat diet (HFD)-induced, obese, atherosclerosis-prone mouse LDLr knockout (KO). These findings are very promising and suggest that fish protein-derived peptides or amino acids may also explain the beneficial effects of dietary fish intake on the MetS, T2D and CVD. Additional studies are required to validate these observations, delineate the mechanisms, and assess their direct impact in human clinical trials.

Subjects will take an oral dose of 15 g of SPF or comparator per day (powder mixed with water) in the first intervention phase (6 weeks), then 7.5 g of SPF or comparator per day (powder mixed with water) in the second intervention phase (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 35 kg/m2
* Waist circumference ≥ 94 cm for men and ≥ 80 cm for women
* Meet at least one of the following criteria:

Plasma TG > 1.35 mmol/L Fasting glycemia ≥ 5,6 mmol/L and ≤ 6,9 mmol/L HbA1c ≥ 5,7% and ≤ 6.4% Insulin concentration > 42 pmol/L

Exclusion Criteria:

* Smoker
* Suffering from any metabolic disorder requiring pharmacological treatment
* Taking any medications or natural health products affecting glucose metabolism or plasma lipid levels
* Use of protein supplements, probiotics supplements or antibiotics within the last 3 months
* Taste aversion for fish/seafood
* Fish-seafood or casein/milk protein or any non-medicinal ingredients allergy
* Lactose intolerance
* Regular alcohol consumption (>2 drinks/d)
* >5% weight loss over the last 3 months
* Major surgery within the last 3 months
* Pregnant and breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Change in hepatic enzymes using blood sampling | Change between the beginning and the end of the intervention (6 weeks)
  Measure hepatic enzymes aspartate aminotransferase (AST), alanine aminotransferase (ALT) and gamma glutamyl transferase (GGT) to test the safety of SPF
Change in renal function using blood sampling | Change between the beginning and the end of the intervention (6 weeks)
  Measure creatinine to test the safety of SPF
Change in complete blood count using blood sampling | Change between the beginning and the end of the intervention (6 weeks)
  Measure of complete blood count to test th safety of SPF
Adverse event and general acceptability evaluated by questionnaires | Change between the beginning and the end of the intervention (6 weeks)
  To test the safety of SPF

SECONDARY OUTCOMES:
Change in lipid profile | Change between the beginning and the end of the intervention (6 weeks)
  Evaluation of plasma triglycerides (TG), Total cholesterol, LDL, HDL, Apolipoprotein B and free fatty acids
Change in glucose metabolism | Change between the beginning and th end of the intervention (6 weeks)
  Evaluation of blood glucose concentration during a 3h oral glucose tolerance test
Change in insulin secretion | Change between the beginning and th end of the intervention (6 weeks)
  Evaluation of blood insulin and C-peptide concentration during a 3h oral glucose tolerance test
Change in blood pressure | Change between the beginning and th end of the intervention (6 weeks)
  Evaluation of systolic and diastolic blood pressure to test metabolic syndrome risk factors
Change in body mass index | Change between the beginning and th end of the intervention (6 weeks)
  Evaluation of BMI by measuring weight and height to test metabolic risk factors
Change in waist circumference | Change between the beginning and th end of the intervention (6 weeks)
  Measure of waist circumference to test metabolic risk factors

CONTACTS AND LOCATIONS:
Locations (1):
- INAF, Université Laval, Québec, Quebec, Canada